CLINICAL TRIAL: NCT02976103
Title: Reduction of Post Mastectomy Pain With the Jacki® Recovery Jacket: Randomized Trial
Brief Title: Reduction of Post Mastectomy Pain With the Jacki® Recovery Jacket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Daisy Foundation (Other)
Responsible Party: Principal Investigator, Donna Berry, PhD, RN, FAAN, AOCN, Donna Berry, PhD, RN, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 16-403
Record Dates: First submitted 2016-11-18; First posted 2016-11-29 (Estimated); Results first posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-02

CONDITIONS: Mastectomy
Keywords: recovery; pain; surgical drains
MeSH Terms: conditions — Pain | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Care (Other): -Standard Care pain medicine/management will be given
  Interventions: Other: Standard Care Pain medicine/management
- JACKI® RECOVERY JACKET + Standard Care (Experimental): * Patient will be encouraged to use the Jacki Recovery Jacket at home
  * Patient will be taught how to tuck the drainage tubes in the jacket pocket
  * Patient will be taught how to un-tuck the drainage tubes from jacket pocket
  * Standard care pain medicine/management will be given
  Interventions: Device: Jacki Recovery jacket; Other: Standard Care Pain medicine/management

INTERVENTIONS:
Device: Jacki Recovery jacket — An outer jacket that holds surgical drains and allows access for blood draws
  Arms: JACKI® RECOVERY JACKET + Standard Care
Other: Standard Care Pain medicine/management — Standard care pain medicine and management in hospitals where the study enrolls

SUMMARY:
This research study is studying a garment called the Jacki® recovery jacket that can be worn after surgery as a possible way to manage pain from surgical drains.

The study intervention involved in this study is:

-"Jacki" recovery jacket

DETAILED DESCRIPTION:
In this research study, the investigators are studying the Jacki, a garment that can be worn post-mastectomy with pockets that hold post-surgical drains. The Jacki was invented by a cancer survivor who leads A Little Easier Recovery®, a non-profit organization in Massachusetts, and may help participants manage the pain of post-surgical drains to increase comfort and ease of daily living. The jacket has not previously been tested in a research study. The investigators are hoping to learn whether the jacket is effective in reducing pain and discomfort from the time participants leave the hospital until they return to have their drains removed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥ 18 years old.
* Patients who speak and understand English.
* Patients who have had mastectomy with reconstructive surgery in one or both breasts.

Exclusion Criteria:

* Co-morbid delirium
* Dementia
* Mental illness, or neurocognitive deficit prohibiting informed consent and/or ability to complete study procedures.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Berry, PhD, RN, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Berry DL, Blonquist TM, Halpenny B, Hong F, Morrison-Ma SC, McCullough MC, Carelli K, Dominici LS, King TA. The Jacki Jacket after mastectomy with reconstruction: a randomized pilot study. Breast Cancer Res Treat. 2020 Jan;179(2):377-385. doi: 10.1007/s10549-019-05465-9. Epub 2019 Oct 14. PMID 31612292

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment dates: 03/09/2017-12/21/2017
Groups:
- JACKI® RECOVERY JACKET + Standard Care: * Patient will be encouraged to use the Jacki Recovery Jacket at home
  * Patient will be taught how to tuck the drainage tubes in the jacket pocket
  * Patient will be taught how to un-tuck the drainage tubes from jacket pocket
  * Standard care pain medicine/management will be given
  Jacki Recovery jacket: An outer jacket that holds surgical drains and allows access for blood draws
  Standard Care Pain medicine/management: Standard care pain medicine and management in hospitals where the study enrolls
Period: Overall Study
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Started | 67 | 72
Completed | 54 (54 participants answered final (T3) questionnaire) | 64 (64 participants answered final (T3 questionnaire))
Not Completed | 13 | 8
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care | Total
Number analyzed (Participants) | 67 | 72 | 139
Age, Continuous [Median (Full Range); unit: years] | 49 [23 to 75] | 47 [25 to 66] | 48 [23 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 72 | 139
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 60 | 67 | 127
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 60 | 62 | 122
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 67 | 72 | 139
Pain Intensity Numeric (0-10) Scale (PINS) [Mean (Standard Deviation); unit: score on a scale] — 1 item (score 0-10); higher score = worse outcome
  score on a scale | 4.7 (2.2) | 4.7 (2.0) | 4.7 (2.1)
Symptom Distress Scale - Pain Frequency [Mean (Standard Deviation); unit: units on a scale] — Population: 1 participant did not provide a response
  units on a scale
    number analyzed (Participants) | 67 | 71 | 138
    (all) | 3.9 (1.0) | 3.8 (1.1) | 3.9 (1.1)
Symptom Distress Scale - Pain Intensity [Mean (Standard Deviation); unit: units on a scale] | 3.0 (1.0) | 2.8 (0.8) | 3.0 (1.0)
PROMIS Pain Intensity Short Form 3a [Mean (Standard Deviation); unit: score on a scale] — 3 items (T score 0-100); higher score = worse outcome Population: 2 participants did not complete the required items to calculate a total score
  score on a scale
    number analyzed (Participants) | 65 | 72 | 137
    (all) | 54.4 (6.7) | 53.7 (5.4) | 54.0 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity (on the 0-10 Pain Intensity Numeric Scale)
Description: Pain Intensity Numeric Scale (0-10)(higher scores = worse outcome)
Time Frame: 1-2 weeks
Population: Standard Care arm (n=54): 52 of 54 participants who answered T3 with a PINS score, plus 2 participants who answered for the same day in their T2 diary Jacki+Standard Care arm (n=68): 64 of 64 participants who answered T3 with a PINS score, plus 4 participants who answered for the same day in their T2 diary
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 68
score on a scale | 1.9 (1.7) | 2.1 (1.9)

2. Secondary Outcome: Symptom Distress Scale - Pain Frequency
Description: 1 item (score range 1-5); higher score = worse outcome
Time Frame: 1-2 weeks
Population: 13 participants in the standard care arm and 8 in the Jacki Jacket arm (total of 21) did not answer the T3 questionnaire or did not answer this item
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 2.9 (1.2) | 2.9 (1.1)

3. Secondary Outcome: Symptom Distress Scale - Pain Intensity
Description: 1 item (score range 1-5); higher score = worse outcome
Time Frame: 1-2 weeks
Population: 14 participants in the standard care arm and 8 in the Jacki Jacket arm (total of 21) did not answer the T3 questionnaire or did not answer this item
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 53 | 64
score on a scale | 2.0 (0.9) | 2.1 (0.9)

4. Secondary Outcome: PROMIS Pain Intensity Scale (Short Form 3a)
Description: 3 items (T score 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Population: 13 participants in the Standard Care arm and 9 in the Jacki Jacket arm (Total of 21) did not provide complete data to calculate this scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 63
score on a scale | 46.8 (7.0) | 46.1 (5.3)

5. Secondary Outcome: PROMIS Pain Interference Scale - Short Form 8a
Description: 8 items (T score 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Population: 13 participants in the Standard Care arm and 10 in the Jacki Jacket arm (total of 23) did not complete answer the T3 questionnaire or did not answer all items required to calculate a score
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 62
score on a scale | 58.9 (8.4) | 59.1 (7.5)

6. Secondary Outcome: EORTC QLQ-C30: Global QOL Scale
Description: 2 items; score range 0-100 (higher score = better outcome)
Time Frame: 1-2 weeks
Population: T3 respondents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 66.0 (17.2) | 64.1 (16.7)

7. Secondary Outcome: EORTC QLQ-C30: Physical Functioning Scale
Description: 5 items; score range 0-100 (higher score = better outcome)
Time Frame: 1-2 weeks
Population: T3 respondents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 53 | 62
score on a scale | 76.3 (23.9) | 71.7 (20.0)

8. Secondary Outcome: EORTC QLQ-C30: Role Functioning Scale
Description: 2 items; score range 0-100 (higher score = better outcome)
Time Frame: 1-2 weeks
Population: T3 respondents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 62
score on a scale | 36.1 (27.2) | 40.3 (24.6)

9. Secondary Outcome: EORTC QLQ-C30: Emotional Functioning Scale
Description: 4 items; score range 0-100 (higher score = better outcome)
Time Frame: 1-2 weeks
Population: T3 respondents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 72.8 (20.1) | 73.3 (21.7)

10. Secondary Outcome: EORTC QLQ-C30: Cognitive Functioning Scale
Description: 2 items; score range 0-100 (higher score = better outcome)
Time Frame: 1-2 weeks
Population: T3 respondents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 84.0 (22.9) | 81.0 (21.6)

11. Secondary Outcome: EORTC QLQ-C30: Social Functioning Scale
Description: 2 items; score range 0-100 (higher score = better outcome)
Time Frame: 1-2 weeks
Population: T3 respondents
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 59.0 (28.7) | 56.5 (26.7)

12. Secondary Outcome: EORTC QLQ-BR23: Body Image Subscale
Description: 4 items (score 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 53 | 64
score on a scale | 56.6 (29.8) | 64.8 (25.0)

13. Secondary Outcome: EORTC QLQ-BR23: Sexual Functioning Subscale
Description: 2 items (range 0-100); higher score = better outcome
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 49 | 57
score on a scale | 18.0 (18.3) | 15.8 (19.0)

14. Secondary Outcome: EORTC QLQ-BR23: Sexual Enjoyment Subscale
Description: 1 item (range 0-100); higher score = better outcome
Time Frame: 1-2 weeks
Population: The majority of respondents skipped this item because they were not sexually active in the time period immediately after surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 17 | 22
score on a scale | 54.9 (35.2) | 57.6 (29.4)

15. Secondary Outcome: EORTC QLQ-BR23: Future Perspective Subscale
Description: 1 item (range 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 49.4 (30.2) | 53.1 (30.1)

16. Secondary Outcome: EORTC QLQ-BR23: Systemic Therapy Side Effects Subscale
Description: 7 items (range 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 13.4 (12.6) | 15.4 (12.8)

17. Secondary Outcome: EORTC QLQ-BR23: Breast Symptoms Subscale
Description: 4 items (range 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 32.8 (21.9) | 31.4 (21.7)

18. Secondary Outcome: EORTC QLQ-BR23: Arm Symptoms Subscale
Description: 3 items (range 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 54 | 64
score on a scale | 30.9 (20.2) | 30.9 (19.8)

19. Secondary Outcome: EORTC QLQ-BR23: Upset by Hair Loss Subscale
Description: 1 item (range 0-100); higher score = worse outcome
Time Frame: 1-2 weeks
Population: Most participants did not answer this item as they had not experienced hair loss (did not receive chemotherapy prior to surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 8 | 11
score on a scale | 25.0 (38.8) | 24.2 (33.6)

20. Secondary Outcome: Pain Patterns At Home: Average Daily Pain Intensity (Daily Diary)
Description: Average 0-10 Pain Intensity Numeric Scale Rating, for 7 days post-discharge, if at least 5 days reported (T2 diary)
Time Frame: 1 week
Population: 16 in Jacki arm and 21 in Standard Care arm did not return T2 diary; 2 in Standard Care arm returned diary with missing data, for a total of 23 missing this measure in Standard Care arm
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 44 | 16
units on a scale | 3.6 [3.0 to 5.0] | 4.4 [2.9 to 5.4]

21. Secondary Outcome: Pain Management At Home: Use of Pain Medication (Daily Diary)
Description: Participant self-report of average daily morphine eqivalent dose taken in first 7 days post-discharge (if at least 5 days reported)
Time Frame: 1-2 weeks
Population: Participants who returned T2 diary with sufficient information on medication usage to calculate a 7-day average morphine equivalent dose
Measure: Median (Inter-Quartile Range); unit: morphine equivalent dose units
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 42 | 52
morphine equivalent dose units | 6.9 [2.3 to 16.1] | 10.7 [2.2 to 28.3]

22. Secondary Outcome: Pain Management At Home: Use of Mastectomy Bra (Daily Diary)
Description: Self-reported proportion of days in the first 7 days post discharge that participant wore a mastectomy bra (if at least 5 days reported)
Time Frame: 1-2 weeks
Population: Participants who returned a T2 diary with sufficient data on wearing a mastectomy bra to calculate a proportion for the first 7 days post-discharge
Measure: Median (Inter-Quartile Range); unit: Proportion of days
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 42 | 52
Proportion of days | 1.0 [0.0 to 1.0] | 1.0 [1.0 to 1.0]

23. Secondary Outcome: Pain Management At Home: Use of Mastectomy Camisole (Daily Diary)
Description: Self-reported proportion of days in the first 7 days post discharge that participant wore a mastectomy camisole (if at least 5 days reported)
Time Frame: 1-2 weeks
Population: Participants who returned a T2 diary with sufficient data on wearing a mastectomy camisole to calculate a proportion for the first 7 days post-discharge
Measure: Median (Inter-Quartile Range); unit: Proportion of days
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 42 | 52
Proportion of days | 0.8 [0.0 to 1.0] | 0.1 [0.0 to 0.9]

24. Secondary Outcome: Patient-Reported Usage of Jacki Recovery Jacket (Daily Diary)
Description: Self-reported proportion of days in the first 7 days post-discharge that participant wore the Jacki recovery jacket at all; no score is better or worse
Time Frame: 1-2 weeks
Population: Summary measure for participants in the Jacki Recovery Jacket + Standard Care arm only. A proportion score was calculated if the measure was reported for at least 5 of the first 7 days post-discharge. Of 73 participants assigned to this arm, 53 returned a T2 diary, and 49 had sufficient data to calculate a proportion score.
Measure: Median (Inter-Quartile Range); unit: Proportion of days
Arm/Group | JACKI® RECOVERY JACKET + Standard Care
Number analyzed (Participants) | 49
Proportion of days | 0.9 [0.6 to 1.0]

ADVERSE EVENTS:
Time Frame: Adverse events were collected only when the participant was on study (usually 1-6 weeks).
Description: Per protocol, adverse events that could reasonably be expected to relate to the NSR device (jacket) included:
  1. Dislodging post-surgical drains, possibly resulting in infection
  2. Becoming over warm or irritating skin
  Data were collected by chart review and patient report either verbally to the study coordinator or on the study diary.
Arm/Group | Standard Care | JACKI® RECOVERY JACKET + Standard Care
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/72
Other Adverse Events (participants affected / at risk) | 0/67 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT02976103/Prot_SAP_000.pdf